CLINICAL TRIAL: NCT00411593
Title: Phase I-II Study of Avastin®+ Bortezomib for Patients With Recurrent or Refractory Non-Squamous NSCLC
Brief Title: Phase I-II for Patients With Recurrent or Refractory Non-small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Patient Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0045
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; NSCLC; Bortezomib; Bevacizumab
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin® + Bortezomib (Experimental): Phase I - 3 * 3 design, enrolling patients to receive Avastin® at a fixed dose of 15 mg/kg every 3 weeks and Bortezomib dosed at 1.6 mg/m2 weekly for 2 weeks out of 3.
  Phase II - The MTD for Bortezomib from the weekly schedule that is chosen will be combined with Avastin® to estimate the rate of progression-free survival.
  Interventions: Drug: Bevacizumab; Drug: Bortezomib

INTERVENTIONS:
Drug: Bevacizumab — 15 g/kg by vein every 3 weeks on day 1 of each cycle.
  Other Names: Avastin; Anti-VEGF Monoclonal Antibody; rhuMAb-VEGF
Drug: Bortezomib — Phase I Starting dose: 1.6 mg/m2 by vein on days 1, 8 of each 3 week cycle.
  Phase II: MTD from Phase I.
  Other Names: Velcade; LDP-341; MLN341; PS-341

SUMMARY:
Primary Objective

The primary objective of this phase I-II study is to evaluate:

* Phase I: Assess the maximum tolerated dose (MTD) of bortezomib in a weekly schedule with bevacizumab given every 3 weeks.
* Phase II: Using the MTD established in phase I, assess efficacy of the combination as indicated by progression-free survival.

Secondary Objectives

The secondary objectives of this study are to evaluate:

* Response rates and duration of response
* 1 year survival
* Overall survival
* Qualitative and quantitative toxicity
* Circulating endothelial cells (CECs) prior to treatment, prior to cycle 2, and/or at the time of progression

DETAILED DESCRIPTION:
Bortezomib is designed to enter cells and interfere with a substance found inside cells that is responsible for allowing cells to divide.

Avastin® is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

If you are found to be eligible to take part in this study, depending on when you enroll, you will be assigned to one of up to 4 treatment groups. There will be 3 participants in each of the first few groups, and an additional 30 participants in the last group. The first few (2 or 3) groups are part of the first phase of the study, and the last group (3rd or 4th) is part of the second phase. All participants will receive the same dose level of Avastin®. The amount of bortezomib you receive will depend on when you enroll in the study. The exact dose of bortezomib that you receive will be based on your height and weight. In the first phase of the study, groups of participants will be assigned to one of 2 bortezomib dose levels. The first group will receive the highest dose. The next groups will receive either that same dose level, or if intolerable side effects occurred, a lower dose level. For the second part of the study, the last group will receive the highest dose level that did not cause intolerable side effects in the other groups.

A cycle of treatment is 3 weeks (21 days). Bortezomib will be given once a week for the first 2 weeks of each cycle. Avastin® will be given every 3 weeks. (On Day 1 of each cycle, you will receive both bortezomib and Avastin®.)

Bortezomib will be injected through a needle in your vein. Each injection will last about 3-5 seconds. After receiving each dose of bortezomib, the clinic staff will check how well you are tolerating the drug. During that time, you will be asked about any side effects you may be experiencing. Your doctor may decrease or pause the dose of bortezomib if you experience certain side effects.

Avastin® will be given as an infusion through a needle in your vein, over 90 minutes. If you tolerate the 90-minute infusion well, the second infusion will be given over 60 minutes. If you tolerate the 60-minute infusion well, all following infusions will be given over 30 minutes. If you do not tolerate the shorter infusion time, future infusion times will be increased until a tolerable level is reached.

Every 3 weeks, you will have a physical exam, including measurement of vital signs and weight. Blood (about 2 teaspoons) will be drawn for routine tests. You will have a performance status evaluation. On Day 8 of each cycle of treatment, blood (about 2 teaspoons) will be drawn for routine tests. The level of protein in your urine will be monitored at least every 6 weeks.

You may continue receiving study treatment for as long as the cancer responds to the treatment or for up to 1 year. Your doctor may decide to take you off this study if you experience intolerable side effects or your health gets worse.

After you have stopped taking the study treatment, you will have a physical exam, including measurement of vital signs. Blood (about 2 teaspoons) will be drawn for routine tests. You will have a performance status evaluation, chest x-ray, and a CT or MRI scan. On an indefinite basis, the study nurse will contact you by telephone from time to time to see how you are doing.

This is an investigational study. Bortezomib has been FDA approved and it is registered in Europe for the treatment of multiple myeloma patients who have received at least one prior therapy. Avastin® has been FDA approved for the treatment of metastatic colorectal cancer and non-small cell lung cancer. However, bortezomib and Avastin® are not FDA-approved for this type of cancer, and they have been authorized for use together in research only. Up to 42 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Female subject is either post-menopausal (Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential) or surgically sterilized or willing to use an acceptable method of birth control (i.e. a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study.
3. All patients must have an Eastern Cooperative Oncology Group (ECOG)Performance Status of 0 - 2
4. Patients must have histologically or cytologically proven selected Stage IIIB (T4 lesion due to malignant pleural or pericardial effusion) or Stage IV advanced non-small cell lung cancer or recurrent disease after previous surgery and/or radiation.
5. No history of or active brain metastases
6. Patients must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI). Measurable disease must be assessed within 28 days prior to registration. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease.
7. Recurrent or progressive cancer can be within a previously radiated site
8. Patients must have received one or two prior systemic therapies, one of which contained a platinum compound. No prior Bortezomib or antiangiogenic agent is permitted. Prior radiation is permitted; however, at least two weeks must have elapsed since the completion of prior radiation therapy and patients must have recovered from all associated toxicities at the time of registration. At least two weeks must have elapsed since surgery (thoracic or other major surgeries) and patients must have recovered from all associated toxicities at the time of registration.
9. Patients must have a serum creatinine </= the institutional upper limit of normal (i.e. 1.5 mg/dL) AND a creatinine clearance >/= 40 cc/min determined by either urine collection and testing or calculation using the following formula: Calculated Creatinine Clearance = (140 - age) * Weight(kg) * (0.85 if female)/ 72 * creatinine (mg/dL)
10. Patients must have an Absolute neutrophil count (ANC)>/= 2,000/µl and platelet count >/= 100,000/µl obtained within 28 days prior to registration. Hemoglobin: >9.0 * 10^9/L
11. Patients must have adequate hepatic function documented by a serum bilirubin </= institutional upper limit of normal (1.0) and liver enzymes (serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT)) </= 3.0 * the institutional upper limit of normal obtained within 28 days prior to registration
12. Peripheral neuropathy, if present, must be < Grade 2 (NCI Common Terminology Criteria for Adverse Events Version 3.0).
13. Patients known to be HIV-positive and taking HAART therapy are not eligible due to possible pharmacokinetic interactions
14. Patients must not be planning to receive any other concomitant anticancer treatment including chemotherapy, radiation therapy, biologic agents or any other investigational drugs
15. Patient must be >/= 18 years of age.
16. Patients must be informed of the investigation nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Patients meeting any of the following exclusion criteria are not to be enrolled in the study. Participation in an experimental drug study within 4 weeks of the first treatment on this trial: Blood pressure > 140/90 mm Hg, History of stroke within 6 months, Clinically significant peripheral vascular disease, Evidence of bleeding diathesis or coagulopathy, Presence of central nervous system or brain metastases
2. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study.
3. Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
4. Urine protein: creatinine ratio >/= 1.0 at screening
5. Serious non-healing wound, ulcer, or bone fracture
6. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class II or heart failure, unstable angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, and ECG abnormality at Screening has to be documented by the investigator as not medically relevant
7. Patients with squamous histology
8. Patients with hematemesis or more than ½ teaspoon of hemoptysis within 6 months of study entry.
9. Patients requiring full dose oral or parenteral anticoagulation.
10. Abdominal fistula, GI perforation, or abdominal abscess within the last 6 months
11. Patient has hypersensitivity to boron or mannitol
12. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women. Patient has received other investigational drugs within 28 days before enrollment
13. Serious medical or psychiatric illness likely to interfere with participation in this clinical study
14. No other prior or concurrent malignancy is allowed except for: non-melanoma skin cancers, in situ cervical cancer, and any cancer from which the patient has been disease-free for 3 years or more.
15. Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including fetal death from the chemotherapeutic agents. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
16. Patients requiring treatment with Nonsteroidal anti-inflammatory drugs (NSAIDS), antiplatelet agents, or aspirin > 325 mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 days
  MTD is defined as the highest dose level in which 6 patients have been treated with 2 patients with dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
  Patients' progression free survival, 1 year survival and overall survival will be assessed. The survival rate for time to event outcome will be estimated by Kaplan-Meier method. All patients will be followed until death.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S. Glisson, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://mdanderson.org